CLINICAL TRIAL: NCT00727480
Title: Finger Imaging and Biometric System
Brief Title: Finger Imaging to Detect Blood Flow in the Fingertips
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer acruing data for this study.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Paul L. Carson Ph.D, Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2002-0535
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Capillary Permeability
Keywords: vascularity; fingertips
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Ultrasound Imaging of fingertips
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound scanning of fingertips for assessment of possible imaging modes with Gray scale ultrasound, color flow vascularity imaging, and color flow vascularity imaging before and after exercise.

SUMMARY:
The purpose of this study is to develop a small, easily used device to detect a person's blood flow in their fingertips.

DETAILED DESCRIPTION:
To develop a hand held touch-pad device for identification of individuals, to help with banking and, possibly for detection of anxiety. This is done by their fingerprint and, other digital anatomy and vascular biometrics.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female who can give informed consent

Exclusion Criteria:

* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2002-09; Primary Completion 2008-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To develop a new type of electronic hand held device, that will demonstrate the image quality comparable to existing devices based on optical techniques. | 2002-2011

CONTACTS AND LOCATIONS:
Overall Officials: Paul L. Carson, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States